CLINICAL TRIAL: NCT00145197
Title: Improving the Delivery of Effective Care to Minorities
Brief Title: Reducing Underuse of Early-Stage Breast Cancer Treatment in Minority Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: GCO 00-0053; 5P01HS010859-05 (AHRQ)
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; adjuvant treatment; racial disparities; Early-Stage Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Improving the Delivery of Effective Care to Minorities (Experimental)
  Interventions: Behavioral: Improving the Delivery of Effective Care to Minorities

INTERVENTIONS:
Behavioral: Improving the Delivery of Effective Care to Minorities — The intervention consists of: a) reminders to prompt surgeons to refer patients for adjuvant treatment, and b) an individual to track referrals for and receipt of adjuvant treatments. We will recruit all physicians who treat patients with early stage breast cancer. Physicians who agree to participate will identify a point person in their office who will inform the research team if the patient has a follow up appointment with radiation or medical oncologists. Following the appointment date, we will contact each office to confirm the patient's visit. If the patient has connected with radiation and/or medical oncologist, we will let the surgeon's office know and stop calling his/her office. However, if the patient has not made the appropriate visits, we will continue to call the surgeon's office every week for a total of 3 calls to let them know that the patient has not connected with the oncologist.

SUMMARY:
The purpose of this study is to determine if a physician-centered intervention will help women with early stage breast cancer receive appropriate treatment.

DETAILED DESCRIPTION:
Efficacious adjuvant treatments such as radiotherapy following breast conserving surgery, and chemo- or hormonal therapy for stage 1b or 2 breast cancer improve disease-free and overall survival. Lower rates of radiotherapy following breast-conserving surgery have been reported among black women. Few data exist about racial disparities in receipt of chemo- or hormonal therapies; however, poorer stage-specific survival rates among blacks and among women with poor or no insurance suggest underuse of these treatments. Despite elimination of racial disparities in rates of mammography screening, the full benefit of screening will not be realized unless underuse of effective treatments for early-stage breast cancer is eliminated. Little is known about reasons for underuse of these treatments or ways to increase treatment rates. Our preliminary work suggests omitted referrals and lack of follow-up tracking account for a majority of underuse particularly among minority patients.

The proposed breast cancer project will measure the extent of underuse of efficacious breast cancer treatments among patients of the hospitals serving East and Central Harlem and other minority communities in lower Manhattan. We will first interview physicians and patients about their reasons for omission of efficacious adjuvant treatments. At the 6 participating hospitals, we will then implement an intervention consisting of: a) computerized reminders to prompt surgeons to refer patients for adjuvant treatment, and b) an individual to track referrals for and receipt of adjuvant treatments. We will assess racial/ethnic differences in rates of underuse and explore racial differences in reasons for underuse.

We will assess the impact of the intervention on reducing underuse of efficacious therapies among 2 years of 695 pre-intervention and 2 years of 695 post-intervention patients. This study will provide new knowledge about racial disparities in treatment for early-stage breast cancer; patient and physician reasons for underuse; and the effectiveness of a simple, sustainable intervention to improve rates of efficacious adjuvant treatments.

ELIGIBILITY:
Inclusion Criteria:

* All patients, who are English or Spanish speaking, with a new primary stage 1 or 2 breast cancer who have undergone either breast conserving surgery or mastectomy and those with tumors > 1 cm or < 1 cm and poorly differentiated
* All surgeons performing breast surgery at the participating hospitals

Exclusion Criteria:

* Patients with dementia or those with a poor prognosis due to end-stage organ failure or other concomitant conditions such as those undergoing treatment for other cancers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1164 (Actual)
Dates: Start 2004-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
initiation and completion of primary treatment | measured 6 months after patient recruitment

SECONDARY OUTCOMES:
adherence | measured at time of patient survey
emotional and health status | measured at time of patient survey
patient satisfaction | measured at time of patient survey
knowledge & beliefs | measured at time of patient survey

CONTACTS AND LOCATIONS:
Overall Officials: Nina Bickell, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States